CLINICAL TRIAL: NCT04927130
Title: An International Multicenter Blind Retrospective Comparative in Vitro Case-controlled Study of the ARNA Breast Liquid Biopsy Test System in Women With Biopsy Confirmed Breast Cancer
Brief Title: Retrospective Comparative in Vitro Case-controlled Study of the Liquid Biopsy Test System in Women With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ARNA Genomics US Inc. (Industry)
Collaborators: BIOMARKER-RU (Unknown)
Responsible Party: Sponsor
Other Study IDs: AB PoC 2021 RUS
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women in age 35 to 65 with confirmed breast cancer
  Interventions: Diagnostic Test: ARNA Breast
- Healthy Volunteers
  Interventions: Diagnostic Test: ARNA Breast

INTERVENTIONS:
Diagnostic Test: ARNA Breast — A specific DNA fragments and globulins will be detected in blood plasma.

SUMMARY:
Proof of Concept retrospective study. Women who have the diagnosis Breast Cancer ( confirmed by biopsy) will donate a blood samples. Tubes with blood will be transferred to the Sponsors Laboratory and ARNA Breast Test will be performed. The result of test will be compared with the biopsy result for each person.

ELIGIBILITY:
Inclusion Criteria:

* Availability of signed and dated informed consent.
* Women from 35 to 65 years old, who are generally healthy, with confirmed breast cancer. Or without any neoplasms in breast (control group)
* Presence of a documented biopsy
* Presence of mammography, ultrasound or MRI of the mammary glands no later than three months.

Exclusion Criteria:

* Pregnancy.
* Any other cancers diagnosed now or previously, with the exception of breast cancer.
* Therapy with cytostatic during the last three months.
* Chemotherapy within the past three months.
* Therapy with hormonal drugs, including all forms of contraceptive drugs.
* Therapy with other prohibited groups of drugs.
* Systolic blood pressure > 180 mm Hg. and / or diastolic blood pressure > 120 mm Hg. with repeated measurements.
* Simultaneous participation in another clinical study.
* Relative affiliation to the clinic, for example, the patient is a close relative of the researcher or a dependent person (for example, a clinic employee or student or a sponsor employee).
* A clinically significant condition or laboratory result that, in the opinion of the investigator, threatens the safety of the test subject, may interfere with assessments, or prevent the completion of the study.
* Failure to cooperate to participate in planned procedures, including the following examples: lack of understanding of language, mental illness, inability to visit the clinic.
* Diseases or conditions that may affect the conduct of the study or the interpretation of the results.
* History of organ transplantation.
* Blood transfusions within the last 6 months.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women of the required age group, in case of breast cancer has been confirmed but not treated, are sent to donate blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-29 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of true positive cases | through study completion, an average of 1 year
  the absolute total number of matches between the results of the test system and histological confirmation of the diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- K+31, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided